CLINICAL TRIAL: NCT01191372
Title: First-in-Human and Proof-of-Mechanism Study of ARC19499 Administered to Hemophilia Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARC19499-001; 2010-020373-17 (EudraCT Number); 271101 (Other: Baxter Healthcare Corporation)
Record Dates: First submitted 2010-08-26; First posted 2010-08-30 (Estimated); Last update posted 2021-05-05 (Actual); Status verified 2021-05

CONDITIONS: Hemophilia
Keywords: Hemophilia A; Hemophilia B; pharmacokinetics; pharmacodynamics; Tissue Factor Pathway Inhibitor
MeSH Terms: conditions — Hemophilia A; Hemophilia B | interventions — ARC19499

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- saline for injection (Placebo Comparator)
  Interventions: Drug: placebo control
- ARC19499 Low Dose (Experimental)
  Interventions: Drug: ARC19499
- ARC19499 Mid Dose (Experimental)
  Interventions: Drug: ARC19499
- ARC19499 High Dose (Experimental)
  Interventions: Drug: ARC19499

INTERVENTIONS:
Drug: placebo control — sterile saline for injection
  Arms: saline for injection
Drug: ARC19499 — Anti-tissue factor pathway inhibitor (TFPI) aptamer
  Arms: ARC19499 High Dose; ARC19499 Low Dose; ARC19499 Mid Dose

SUMMARY:
The purpose of this study is to examine the safety, tolerability and the way the body handles various single and multiple doses of ARC19499 in patients with hemophilia.

ELIGIBILITY:
Inclusion Criteria:

Adult male patients ≥18 to ≤75 years of age.

* Hemophilia of any type or severity.
* Patients who are negative for hepatitis B surface antigen (HBsAg), and human immunodeficiency virus (HIV) I and II antibody tests at screening.
* Male patients who, with their partners, are willing to use 2 effective, methods of contraception (i.e., for both self and partner) throughout the study and for at least 3 months after discontinuation of study drug treatment.
* All patients must be capable of understanding and complying with the protocol and must have signed the informed consent document.

Exclusion Criteria:

* Female patients;
* If on a prophylactic coagulation factor concentrate regimen, inability or unwillingness to discontinue prophylaxis during participation in this study.
* Existence of other co-existing bleeding disorder (e.g., von Willebrand Disease).
* Medical history of venous or arterial thromboembolism.
* Scheduled for elective surgical procedure during the conduct of this study.
* Use of an investigational drug within 30 days of study entry.
* Transaminase values > 3 x upper limit of normal (ULN) at time of screening.
* Haemoglobin <12.0 g/dL.
* Participants who, in the opinion of the Investigator, have a significant infection or known inflammatory process on screening.
* Participants who have a clinically relevant history or presence of respiratory, gastrointestinal, renal, hepatic, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, connective tissue diseases or disorders.
* Any medical condition the investigator believes would place the patient at increased risk as a result of participation in the study e.g. history of thromboembolic disease or stroke.
* Any medication the investigator considers may increase the risk of adverse effects during the study.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2010-09-15 (Actual); Primary Completion 2011-12-28 (Actual); Study Completion 2011-12-28 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) of ARC19499 | 2 weeks
  The PK profile of ARC19499 administered by single and multiple subcutaneous injections will be characterized. The bioavailability of subcutaneously injected ARC19499 relative to that of intravenously infused ARC19499 will be determined.

SECONDARY OUTCOMES:
Coagulation system pharmacodynamic (PD) effects of ARC19499. | 2 weeks
  The PD profile of ARC19499 with respect to the kinetics of thrombin generation and clot formation will be characterized.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- London, United Kingdom